CLINICAL TRIAL: NCT01296490
Title: Assessing Physical Fitness Effect on the Different Oxidative Stress Measurements, at Rest and After Acute Exercise
Brief Title: Physical Fitness Effect on the Different Oxidative Stress Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wingate Institute (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Eyal Shargal, Director, Sports medicine and research center, Wingate Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Wingate 05
Record Dates: First submitted 2011-02-03; First posted 2011-02-15 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Oxidative Stress
Keywords: oxidative stress, physical exercise, fitness level
MeSH Terms: conditions — Motor Activity | interventions — Exercise Test; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress test (Experimental): The men will run on a treadmill for 10 minutes until exhaustion. Blood will be drawn before, 5 minutes after and an hour after the test.
  Interventions: Other: Stress test

INTERVENTIONS:
Other: Stress test — Stress test while running on a treadmill until exhaustion for 8-12 minutes. Blood will be drawn before, 5 minutes after and an hour after the test.
  Other Names: blood test

SUMMARY:
Physical exercise has many benefits, although it might also have negative impact on the body, which changes in accordance with training level, length of workout, age of subject and their fitness level. These outcomes are governed by complex biological processes, from which Reactive Oxygen Substances (ROS) are considered the most prominent ones during exercise activity. These substances harm muscle activity, and might cause other health related damage by influencing other pathways that engage with free radicals. Excess of ROS, is expressed as Oxidative Stress (OS), pathogenic process activation and aging. With this in mind, it is important to remember that ROS are essential to the investigators bodies as well, especially in gene regulation. Thus they influence proteins that are important for proper muscle function and the immune system.

Physical exercise induces changes in low molecular weight antioxidants, and in antioxidant enzymes. According to results that were published in the literature, no universal conclusion can be made regarding physical exercise effect on antioxidants activity. These contradictions might be attributed to the difference between the methods that were used, and their quality.

Paradoxically, physical exercise has the same effect on ROS inducement in skeletal muscle fibers as does not using the muscles for a long period of time (especially as a result of handicap). It is well known that physical exercise effect oxidative stress and antioxidant. Due to the doubts that rise from the literature, the investigators think that it is important to test physical fitness effect on oxidative stress biological markers, using various high quality methods, on the same population.

The investigators will test healthy men, 20-35 years of age, none smokers with 6-24% fat, who do not take vitamins or supplements. The men will run on a treadmill for 10 minutes to exhaustion, and blood will be taken before the test, 5 minutes after the test, and an hour after the test (checking recovery).

DETAILED DESCRIPTION:
Things the investigators will measure:

1. Filling out a physical fitness, and overall health form, that indicates all fitness activity in the past 3 years, and vitamins and supplements that are being taken.
2. Fat percentage
3. VO2 max
4. Oxidants and antioxidants activity: Super oxide dismutase, Catalase, GSH/GSSG, Glutathione peroxide, Glutathione reductase, LDL, conjugated dienes, Plasma malondialdehyde. Measurements will be taken before the test, 5 minutes after the test and an hour after the test.

Work plan:

50 men, at the ages of 20-35 will be recruited. The participants will fill out a form that indicates their physical activity in the past 3 years, as well as their vitamin and supplements intake.

The men will run on a treadmill for 10 minutes until exhaustion.

Blood will be drawn before, 5 minutes after and an hour after the test. Oxidative stress will be measured according to the following parameters:

* 10 ml of blood in citrate tube will be centrifuged and analyzed for: Super oxide dismutase, Catalase, GSH/GSSG, Glutathione peroxide, Glutathione reductase.
* 2 ml of blood with no coagulating factors will be centrifuged and analyzed for: LDL, conjugated dienes, Plasma malondialdehyde (TBARS).

Clinical research:

Participants will run on a treadmill for 10 minutes until exhaustion. The men will be divided into 5 groups according to their VO2 max, comparing the oxidants and antioxidants activity between the groups.

Checking the oxidative stress and VO2 dependency (VO2 is an index for physical fitness).

Age: 20-35 Sex: Men Inclusion criteria: Healthy men, 2-35 years of age, with 6-24% body fat. Exclusion criteria: Smokers, and people who use vitamins and supplements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* 20-35 years of age, with 6-24% body fat.

Exclusion Criteria:

* Smokers and subjects who use vitamins and supplements

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Higher increase in oxidative stress inducing factors, and antioxidants in men with lower physical fitness compared with men with higher physical fitness. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dov Lichtenberg, PhD, Study Chair — Tel Aviv University
Locations (1):
- Wingate Institute, Netanya, Israel